CLINICAL TRIAL: NCT01059487
Title: Bringing Acute and Wellness Care to Underserved Populations Using Traditional Chinese Medicine: A Pragmatic Clinical Trial Using Quality of Life Measures in a Community Health Care Setting
Brief Title: Bringing Acute and Wellness Care to Underserved Populations Using Traditional Chinese Medicine
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chicago College of Oriental Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); QualityMetrics (Industry); Inspire Tech Group (Unknown)
Responsible Party: Jeannette Hoyt/Executive Director, Chicago College of Oriental Medicine, Inc. dba Chicago College of Asian Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10-003 CEG; GRANT10504752 (Other: Agency for Health Care Research and Quality)
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Pain Management; Traditional Chinese Medicine
Keywords: Traditional Chinese Medicine; Acupuncture
MeSH Terms: conditions — Agnosia | interventions — Medicine, Chinese Traditional; Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Traditional Chinese Medicine (Other): Assessing efficacy of treating subjects/patients with Traditional Chinese Medicine (TCM) by administering SF-36v2 and PIQ-6 surveys to subjects/patients to create a baseline and then re-assessing quality of life achieved through TCM treatments by administering follow-up SF-12v2 and PIQ-6 surveys every four weeks
  Interventions: Other: Traditional Chinese Medicine

INTERVENTIONS:
Other: Traditional Chinese Medicine — Traditional Chinese Medicine includes acupuncture, herbal, tuina and other accessory techniques
  Other Names: Acupuncture; Tuina; Herbs; Moxabustion

SUMMARY:
At a time when there is so much focus in the United States on reducing the cost of health care delivery while maximizing the effectiveness of health care performance, Traditional Chinese Medicine (acupuncture, herbal treatment, and accessory techniques) offers decision makers a tantalizing option. Traditional Chinese Medicine differs from its biomedical counterpart in that it is highly portable, inexpensive to administer, relies on a conversational diagnostic inquiry system to arrive at differential diagnosis for its patients, and has very few reported side effects associated with treatment. The World Health Organization cites acupuncture has a proven and effective treatment for 28 diseases/disorders including stroke, pain management issues and rheumatoid arthritis; the WHO lists another over 65 diseases for which the therapeutic effect of acupuncture has been shown but for which further proof is needed including alcohol dependence, cancer pain and diabetes mellitus. With the completion of this pragmatic clinical trial and introduction of the Constant Care method of health care delivery to underserved communities on Chicago's south side, the investigators can both utilize an effective plan of health care delivery, advance the research needed to effectively utilize Traditional Chinese Medicine as a low cost therapeutic option in this country, and successfully treat disenfranchised populations that have been traditionally overlooked and that deserve a better health and wellness care future.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 21 and over

Exclusion Criteria:

* Children
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
QualityMetric SF36v-2 Quality of Life | Every four weeks

SECONDARY OUTCOMES:
QualityMetric PIQ-6 | Every four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago College of Oriental Medicine, Inc. dba Chicago College of Asian Medicine, Chicago, Illinois, United States